CLINICAL TRIAL: NCT06375005
Title: The Efficacy and Safety of Telitacicept in the Treatment of Early Diffuse Cutaneous Systemic Sclerosis: a Multicenter, Open-label, Randomized Controlled Study
Brief Title: Efficacy and Safety of Telitacicept in the Treatment of Systemic Sclerosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0381
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-03

CONDITIONS: Diffuse Cutaneous Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — telitacicept; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mycophenolate Mofetil + Telitacicept (Experimental): All patients who enroll in this trial will receive mycophenolate mofetil (MMF), which is a drug commonly given to patients with systemic sclerosis in clinical practice. Participants will be treated with MMF 0.5g twice a day for 48 weeks. Telitacicept will be subcutaneously injected at a dose of 160mg per week, lasting for 48 weeks.
  Interventions: Drug: Telitacicept; Drug: Mycophenolate Mofetil
- Mycophenolate Mofetil (Active Comparator): Participants will be treated with MMF 0.5g twice a day for 48 weeks.
  Interventions: Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Telitacicept — Telitacicept is fusion protein comprising a recombinant transmembrane activator and calcium modulator and cyclophilin ligand interactor (TACI) receptor fused to the fragment crystallizable (Fc) domain of human immunoglobulin G (IgG). Telitacicept binds to and neutralizes the activity of two cell-signalling molecules, B-lymphocyte stimulator (BLyS) and a proliferation-inducing ligand (APRIL), thereby suppressing the development and survival of plasma cells and mature B cells. Telitacicept will be subcutaneously injected at a dose of 160mg per week, lasting for 48 weeks.
  Other Names: Taiai for commercial name
  Arms: Mycophenolate Mofetil + Telitacicept
Drug: Mycophenolate Mofetil — All patients will receive background therapy with Mycophenolate Mofetil (MMF), administered orally at a dose of 0.5g twice daily for 48 weeks.
  Other Names: MMF

SUMMARY:
This study is a prospective, open-label, randomized, controlled, multi-center clinical trial. The aim of this study is to investigate the efficacy and safety of Telitacicept in adults with early diffuse cutaneous systemic sclerosis (dcSSc), with Mycophenolate Mofetil (MMF) administered as a background treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18-70 years old.
* Systemic sclerosis, as defined by ACR/EULAR (American College of Rheumatology/European League Against Rheumatism) 2013 criteria.
* dcSSc (diffuse cutaneous systemic sclerosis) according to the LeRoy criteria.
* Disease duration of ≤ 18 months (defined as time from the first non-Raynaud's phenomenon manifestation).
* ≥ 10 mRSS units at the screening visit.
* Negative serum pregnancy test in a woman of childbearing potential at the screening visit.
* Ability to render informed consent in accordance with institutional guidelines.

Exclusion Criteria:

* Limited scleroderma.
* Disease duration of greater than 3 years.
* Rheumatic autoimmune disease other than SSc.
* Systemic sclerosis-like illness associated with environmental agents such as vinyl chloride, or bleomycin.
* Any prior history of renal crisis.
* Intermediate- or high-risk pulmonary arterial hypertension.
* Pulmonary disease with FVC < 50% of predicted or DLCO (hemoglobin-corrected) < 40% of predicted at screening or requires oxygen therapy.
* Underwent major surgery within 8 weeks prior to randomization or planned major surgery during the trial period.
* Use of immunosuppressive therapies, including methotrexate, azathioprine, hydroxychloroquine, leflunomide, tacrolimus, sirolimus, and mycophenolate mofetil within 4 weeks prior to randomization, and cyclophosphamide within 3 months prior to randomization.
* Use of other anti-fibrotic agents, including colchicine, D-penicillamine, thalidomide, nintedanib, pirfenidone, tyrosine kinase inhibitors (imatinib, nilotinib, dasatinib) within 4 weeks prior to randomization.
* Use of corticosteroids at doses exceeding the equivalent of prednisone 10 mg daily, or intravenous and intramuscular corticosteroid injections within 4 weeks prior to randomization.
* Use of Intravenous Immunoglobulin (IVIG) within 12 weeks within 4 weeks prior to randomization.
* Prior use of belimumab, rituximab, or other B-Cell depleting therapies ever.
* Use of other biologics or small molecule targeted therapies, including anakinra within 1 week prior to randomization, ixekizumab within 2 weeks prior to randomization, and infliximab, certolizumab pegol, golimumab, adalimumab, abatacept, tocilizumab within 8 weeks prior to randomization, and janus kinase inhibitors within 2 weeks prior to randomization.
* Prior use of other cell depletion therapies.
* Concurrent serious medical condition which in the opinion of the investigator makes the patient inappropriate for this study such as severe central nervous system disease，severe heart failure, arrhythmia, unstable atherosclerotic cardiovascular disease, severe GI involvement, severe hypertension or severe diabetes.
* Abnormal results in hepatitis B or hepatitis C testing indicating active or chronic infection.
* Active tuberculosis (TB) or latent TB infection.
* Seropositive for human immunodeficiency virus (HIV) or known history of HIV infection.
* Known active bacterial, viral, fungal, mycobacterial, or other infection，including major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening, or oral antibiotics within 2 weeks prior to screening.
* Primary or secondary immunodeficiency.
* IgA deficiency (<10 mg/dL) or IgG deficiency (<400 mg/dL).
* Participation in another clinical research study involving the evaluation of another investigational drug within 3 months of entry into this study.
* Any of the following at the screening visit: Hemoglobin <8.0 g/dL; WBC <3 x 10^9/L; Neutrophil <1.5 x 10^9/L; platelets <75 x 10^9/L; serum ALT or AST > 1.5 x ULN; TBil > ULN; eGFR < 40mL/min/1.73m^2.
* Malignant disease within 5 years prior to screening, with the exception of excised/cured local basal or squamous cell carcinoma of the skin or carcinoma in situ of the uterine cervix;
* Immunization with a live/attenuated vaccine within 4 weeks prior to randomization.
* Pregnant or breast feeding women or women of childbearing potential not willing to use adequate contraception.
* History of allergic or anaphylactic reactions to human, humanized, or murine monoclonal antibodies.
* Immunization with a live/attenuated vaccine within 4 weeks prior to randomization.
* Patients anticipated to be non-compliant with the protocol requirements or expected not to complete the trial as planned (e.g., those with psychiatric disorders, history of alcohol abuse, drug abuse, or substance misuse).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2027-01-06 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Modified Rodnan Skin Score (mRSS) at Week 48 | Baseline, Week 48
  Skin thickness was assessed by the mRSS. The mRSS was rated with scores ranging from 0 (normal) to 3 (severe skin thickening) across 17 different sites. The total score was the sum of the individual skin scores in the 17 body areas (e.g., face, hands, fingers; proximal area of the arms, distal area of the arms, thorax, abdomen; proximal area of the legs, and distal area of the legs, feet), giving a range of 0-51 units and had been validated for participants with systemic sclerosis (SSc). A negative change from baseline showed improvement.
Percentage of Participants With Treatment-related Adverse Events (AEs) and Serious Adverse Events (SAEs) | Week 52
  An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

SECONDARY OUTCOMES:
Change From Baseline in Modified Rodnan Skin Score (mRSS) at Week 24 | Baseline, Week 24
  Skin thickness was assessed by the mRSS. The mRSS was rated with scores ranging from 0 (normal) to 3 (severe skin thickening) across 17 different sites. The total score was the sum of the individual skin scores in the 17 body areas (e.g., face, hands, fingers; proximal area of the arms, distal area of the arms, thorax, abdomen; proximal area of the legs, and distal area of the legs, feet), giving a range of 0-51 units and had been validated for participants with systemic sclerosis (SSc). A negative change from baseline showed improvement.
Percentage of Participants Who Improved in Modified Rodnan Skin Score (mRSS) by ≥20%, ≥40%, ≥60% From Baseline to Week 24 and Week 48 | Baseline, Week 24 and 48
  Skin thickness was assessed by the mRSS. The mRSS was rated with scores ranging from 0 (normal) to 3 (severe skin thickening) across 17 different sites. The total score was the sum of the individual skin scores in the 17 body areas (e.g., face, hands, fingers; proximal area of the arms, distal area of the arms, thorax, abdomen; proximal area of the legs, and distal area of the legs, feet), giving a range of 0-51 units and had been validated for participants with systemic sclerosis (SSc). A negative change from baseline showed improvement. Percentage of participants who achieved improvement in mRSS by ≥20%, ≥40%, ≥60% from baseline to week 24 and week 48 were reported.
American College of Rheumatology Composite Response Index for Systemic Sclerosis (ACR-CRISS) and Revised ACR-CRISS at Week 24 and 48 | Week 24 and 48
  CRISS forms a composite response index consisting of SSc-related organ involvement and the following five variables: mRSS, FVC percent predicted, physician's and patient's global assessments, and HAQ-DI score. The resulting index is a 2-step process that captures clinically meaningful worsening of internal organ involvement and the core variables that show change.
Change From Baseline in Forced Vital Capacity (FVC) Percent Predicted at Week 24 and Week 48 | Week 24 and 48
  FVC is pulmonary function test and will be conducted as per the study Pulmonary Function Manual, which is based on the American Thoracic Society/European Respiratory Society (ATS/ERS) Consensus Statement. FVC is the maximum amount of air exhaled from the lungs after taking the deepest breath possible. Negative change in FVC percent predicted indicates worsening.
Change From Baseline in Diffusing Capacity of the Lungs for Carbon Monoxide (DLCO) Percent Predicted (Corrected For Hemoglobin) at Week 24 and Week 48 | Week 24 and 48
  Diffusing capacity of the lungs for carbon monoxide (DLCO) measures how much oxygen travels from the alveoli of the lungs to the blood stream. It is used to determine the severity of lung disease. DLCO for a given individual is compared to reference or predicted values.
Change From Baseline in Patient's Global Assessment at Week 24 and Week 48 | Baseline, Week 24 and 48
  Patient global assessment for overall disease represents the patient's assessment of the patient's global scleroderma on a 0 (excellent) -10 (extremely poor) Likert scale. Higher score means worse outcome.
Change From Baseline in Physician's Global Assessment at Week 24 and Week 48 | Baseline, Week 24 and 48
  This assessment represents the physician's assessment of the patient's current disease activity on a 0 (excellent) -10 (extremely poor) Likert scale. Higher score means worse outcome.
Change From Baseline in Short Form-36 (SF-36) Questionnaire at Week 24 and Week 48 | Baseline, Week 24 and 48
  The Short Form 36 (SF-36) is a validated 36 item questionnaire which measures quality of life across eight domains: physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, general health.
Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) Score at Week 24 and Week 48 | Baseline, Week 24 and 48
  The HAQ-DI is a composite measure from which a 'Standard Disability Index' score can be computed to assess a patient's disability level. Generally, a score of 0-1 represents mild to moderate difficulty, 1-2 moderate to severe disability and 2-3 severe to very severe disability. The HAQ-DI comprises 20 items that assess patient abilities across 8 functional activities: dressing, rising, eating, walking, hygiene, reach, grip, and usual activities. Each item is rated on a 4-point scale: 0=Without ANY difficulty, 1=With SOME difficulty, 2=With MUCH difficulty, 3=UNABLE to do. The 8 scores of the 8 sections are summed and divided by 8. In the event that one section is not completed by a subject then the summed score would be divided by 7. The final overall HAQ-DI score ranges from 0 to 3 and positive change indicates worse health-related quality of life (HRQoL).
Change From Baseline in Physical Function Assessed by Scleroderma Health Assessment Questionnaire Disability Index (SHAQ-DI) at Week 24 and Week 48 | Baseline, Week 24 and 48
  SHAQ-DI assessed five scleroderma-specific visual analogue scale (VAS) items to explore the impact of participant's disease. These items were developed to measure the effect of scleroderma on five elements of disease that could have a great impact on a participant's daily activities. Each VAS item was rated separately (0-100 millimeters [mm]), with higher scores indicating more severe disease. The five items were: 1) intestinal disease, 2) breathing problem, 3) Raynaud syndrome, 4) finger ulcers, and 5) overall disease.
Change From Baseline in Tender Joint Counts at Week 24 and Week 48 | Baseline, Week 24 and 48
  28 joints are assessed for tenderness (positive or negative). The number of tender joint counts ranges from 0 to 28. A higher number indicates worse outcome.
Change From Baseline in Swollen Joint Counts at Week 24 and Week 48 | Baseline, Week 24 and 48
  28 joints are assessed for swelling (positive or negative). The number of swollen joint count ranges from 0 to 28. A higher number indicates worse outcome.
Change From Baseline in Digital Ulcer Counts at Week 24 and Week 48 | Baseline, Week 24 and 48
  Digital ulcers refer to lesions (on the finger or distal to the metacarpophalangeal joint) with loss of surface epithelisation and a visually discernible depth.

CONTACTS AND LOCATIONS:
Overall Officials: JING XUE, PhD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (9):
- China (9):
  - Affiliated Hospital of Yangzhou University, Yangzhou, Jiangsu
  - Huashan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University School Of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Changxing People's Hospital, Huzhou, Zhejiang
  - The First Hospital of Jiaxing, Jiaxing, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang